CLINICAL TRIAL: NCT05629091
Title: A Randomised, Open-label Clinical Investigation of Clinical Performance and Safety of the Nanofibrillar Cellulose Wound Dressing FibDex in Paediatric and Adult Patients With Superficial Dermal Burns
Brief Title: An Investigation of Performance and Safety of the Wound Dressing FibDex in Patients With Superficial Dermal Burns
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: UPM Kymmene Oyj announced on April 2, 2025, the closure of Biomedicals business. As a result, FibDex manufacturing and sales will discontinue. The premature termination is due to business decision, not related to any safety concerns of FibDex.
Sponsor: UPM-Kymmene Corporation (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fibdex 1-2022
Record Dates: First submitted 2022-10-12; First posted 2022-11-29 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FibDex (Experimental): FibDex® is a CE-marked NFC wound dressing intended to come into contact with injured skin and specifically split-thickness skin graft wounds, which have breached the dermis.
  Interventions: Device: FibDex
- Epicite hydro (Active Comparator): Epicitehydro is composed of biotechnology derived cellulose and is indicated for treatment of superficial and deep partial thermal and chemical burn wounds (1st and 2nd degree), scalds, skin graft donor sites, abrasions and lacerations
  Interventions: Device: Epicite hydro
- Epiprotect (Active Comparator): Epiprotect is composed of biosynthetic cellulose. It contains a minimum of 95% isotonic saline solution. Epiprotect is intended for treatment of partial thickness wounds. It can also be used as a temporary coverage for full thickness wounds prior to transplantation or other surgical intervention.
  Interventions: Device: Epiprotect

INTERVENTIONS:
Device: FibDex — Nanofibrillar cellulose wound dressing
  Arms: FibDex
Device: Epicite hydro — Wound dressing
  Arms: Epicite hydro
Device: Epiprotect — Wound dressing
  Arms: Epiprotect

SUMMARY:
This is a prospective, randomised, open-label, within-patient controlled, non-inferiority clinical investigation of the nanofibrillar cellulose (NFC) wound dressing FibDex® for treatment of superficial dermal burns in paediatric and adult patients. The clinical performance and safety of FibDex® will be compared to Epicitehydro (QRSKIN GmbH, Würzburg, Germany) and Epiprotect® (S2Medical AB, Linköping, Sweden). Epicitehydro is considered to be the primary comparator. The investigation will be conducted at 2 clinical research sites in Sweden.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent (by the patient and/or the patient's parent[s]/legal guardian[s] as applicable).
2. Patient with superficial dermal burn wound(s) (class II/A) ≤36h as assessed by the Investigator.
3. Patient at least 1 year old.
4. Patient who has at least 3 superficial dermal burn wounds on anatomically equivalent areas or a superficial dermal burn large enough to allow a lateral comparison.
5. Wound area at least 50 cm2 (per wound, if 3 separate wounds) or at least 150 cm2 (if single wound) as judged by the Investigator.

Exclusion Criteria:

1. Patient hyper-sensitive or allergic to, or have had a hypersensitivity/allergic reaction to, any of the dressing components.
2. Pregnant or breast-feeding female.
3. Patient with chemically or electrically induced burns.
4. Other non-burn wound in target wound area.
5. Not suitable for inclusion according to the Investigator.
6. Cognitive dysfunction or psychiatric history (Investigator's discretion).
7. Chronic or presently active skin condition that is judged as interfering with normal wound healing process (Investigator's discretion)
8. Target burns on sensitive skin areas, such as the facial or genital area.
9. Inability or unwillingness of participant or parent(s)/legal guardian(s) to give written informed consent.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-08-12 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of FibDex® compared to Epicitehydro in terms of time to clinical wound healing (days) defined as no need of any dressing (inner or outer) | Within 2 to 3 weeks (until the wound has healed)
  At each clinical visit, the Investigator or delegate will assess and record in the eCRF if the inner dressing(s) has detached and judge whether or not there is a need for outer dressing.

SECONDARY OUTCOMES:
Non-inferiority of FibDex® compared to Epiprotect® in terms of time to clinical wound healing (days) defined as no need of any dressing (inner or outer). | Within 2 to 3 weeks (until the wound has healed)
  At each clinical visit, the Investigator or delegate will assess and record in the eCRF if the inner dressing(s) has detached and judge whether or not there is a need for outer dressing.
Non-inferiority FibDex® compared to Epicitehydro and Epiprotect®, respectively, in terms of re-epithelialisation of the initial wound area over time | Within 2 to 3 weeks (until the wound has healed)
  Percentage of re-epithelialisation will be evaluated by visual observation by the Investigator or delegate and classified according following categories: <50%, 50-75%, 76-90%, 90-95% and 96-100%.
Evaluate degree of experienced pain | Within 2 to 3 weeks (until the wound has healed)
  On Day 1, pain will be measured before application of FibDex® and the comparators and after outer layer dressing application. On the subsequent visits, pain will be measured before (background pain) and after (procedural pain) outer layer dressing change during the wound healing period. Patients aged ≥8 years will rate subjective pain using a Numeric Pain Rating Scale (NPRS) 0-10 (0 representing no pain and 10 representing the worst possible pain). Patients aged 4 to 7 years will rate pain using The Faces Pain Scale 0-10 (0 representing no pain and 10 representing very much pain). The Faces, Legs, Activity, Cry, Consolability (FLACC) 0-10 (0 is relaxed and comfortable and 7-10 is severe pain or discomfort or both) behavioural measurement will be used for assessment of pain in patients aged ≤3 years.
Assess clinical performance in terms of number of wound infections | Within 2 to 3 weeks (until the wound has healed)
  The burn will be diagnosed with wound infection if at least 2 of the criteria based on the definition of burn wound infection stated by the American Burn Association, are fulfilled.
Need for surgical intervention | Within 2 to 3 weeks (until the wound has healed)
  If wounds, during subsequent dressing changes and assessments, is judged as not progressing in a favourable direction, or if time from trauma approaches/exceeds 2 to 3 weeks, surgical intervention should be considered.
Assess clinical performance in terms of length of stay (days) at hospital | Within 2 to 3 weeks (until the wound has healed)
  All patients hospitalised for their burns will be monitored by a research nurse. The day of discharge will be recorded in the eCRF. Any readmission after the initial discharge will also be noted in the eCRF and included in the total length of stay.
Assess clinical performance in terms of number of outer layer dressing changes | Within 2 to 3 weeks (until the wound has healed)
  Outer dressings will be changed at each visit (from Visit 3 and onwards) if deemed appropriate by the Investigator
Evaluate scar quality | 3, 6 and 12 months post burn
  Burn scar outcome will be evaluated using the Patient and Observer Scar Assessment Scale (POSAS). For both the patient and the observer, the score for each item is added (1 - 10 where 10 indicates the worst imaginable sensation or scar and 1 corresponds to normal skin. Moreover, observer scale nominal variables, such as type of pigmentation, may be recorded in category boxes in addition to the 10 point scale. Lastly, the patient and observer score their "Overall Opinion" of the scar compared to normal skin with the same 10 point scale, where 1 is normal skin and 10 is the most markedly different scar.
Monitor Adverse Events (AEs) | Within 2 to 3 weeks (until the wound has healed)
  Frequency, intensity and seriousness of AEs
Monitor Device Deficiencies (DDs) | Within 2 to 3 weeks (until the wound has healed)
  Frequency and nature of DDs

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Huss, Principal Investigator — Burn Centre, Uppsala University Hospital
Locations (1):
- Burn Centre, Uppsala University Hospital, Uppsala, Sweden